CLINICAL TRIAL: NCT05333848
Title: Effects of Internet-based Storytelling Programs in Reducing Mental Illness Stigma With Mediation by Interactivity and Stigma Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hiu Ching Tiffany Fong, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: dre20024
Record Dates: First submitted 2022-03-31; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: COMBO Condition; STIGMA Condition; INTERACT Condition; CONTROL Condition
Keywords: mental illness stigma; Internet-based; interactivity; storytelling; social distance; microaggression
MeSH Terms: conditions — Microaggression

STUDY DESIGN:
Intervention Model Description: A 2x2 factorial design randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COMBO condition (Experimental): An interactive stigma content website.
  Interventions: Behavioral: Internet-based storytelling programs with interactivity and stigma content
- STIGMA condition (Experimental): A non-interactive stigma content website.
  Interventions: Behavioral: Internet-based storytelling programs with stigma content only
- INTERACT condition (Experimental): An interactive non-stigma content website.
  Interventions: Behavioral: Internet-based storytelling programs with interactivity only
- CONTROL condition (Placebo Comparator): A non-interactive non-stigma content website.
  Interventions: Behavioral: Internet-based storytelling programs with no interactivity and no stigma content

INTERVENTIONS:
Behavioral: Internet-based storytelling programs with interactivity and stigma content — Participants viewed an interactive stigma content website. Within 10 minutes post-experiment, participants completed the post-experiment questionnaire. One week after the experiment, participants completed the follow-up questionnaire.
  Arms: COMBO condition
Behavioral: Internet-based storytelling programs with stigma content only — Participants viewed a non-interactive stigma content website. Within 10 minutes post-experiment, participants completed the post-experiment questionnaire. One week after the experiment, participants completed the follow-up questionnaire.
  Arms: STIGMA condition
Behavioral: Internet-based storytelling programs with interactivity only — Participants viewed an interactive non-stigma content website. Within 10 minutes post-experiment, participants completed the post-experiment questionnaire. One week after the experiment, participants completed the follow-up questionnaire.
  Arms: INTERACT condition
Behavioral: Internet-based storytelling programs with no interactivity and no stigma content — Participants viewed a non-interactive non-stigma content website. Within 10 minutes post-experiment, participants completed the post-experiment questionnaire. One week after the experiment, participants completed the follow-up questionnaire.
  Arms: CONTROL condition

SUMMARY:
Mental illness stigma has been a concerning issue globally due to its adverse effects on the recovery of people with mental illness and may delay help-seeking for mental health out of the concern of being stigmatized. With technological advancement, Internet-based mental health stigma reduction interventions have been developed to combat mental illness stigma and the effects have been promising.

The present study aimed to examine the differential effects of Internet-based storytelling programs varied on level of interactivity and stigma content in reducing mental illness stigma.

In the present study, the investigator hypothesized that an Internet-based storytelling program with a combination of interactivity and stigma content would lead to the most significant reduction in public stigma, microaggression, and social distance from people with mental illnesses, followed by Internet-based storytelling program with stigma content-only and interactivity-only, compared with control. Secondly, the investigator hypothesized that the effects observed in stigma reduction would be mediated by perceived autonomy and immersiveness due to the presence of interactivity.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* able to read and understand Chinese

Exclusion Criteria:

* less than 18 years of age
* unable to read or understand Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2020-12-27 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Public Stigma towards People with Mental Illness within 10 minutes post-experiment, and at 1-week follow-up | baseline, within 10 minutes post-experiment, and 1-week follow-up
  The 21-item Public Stigma Scale-Mental Illness-Short Version was used to assess mental illness public stigma and personal advocacy. Each item was rated on a 6-point Likert scale from 1 (strongly disagree) to 6 (strongly agree). Reverse scoring was done for personal advocacy items. Higher scores indicated a higher level of public stigma towards people with mental illness.
Change from Baseline Microaggression within 10 minutes post-experiment, and at 1-week follow-up | baseline, within 10 minutes post-experiment, and 1-week follow-up
  Microaggression was measured by the 17-item Mental Illness Microaggressions Scale, which covers assumption of inferiority, patronization, and fear of mental illness. Each item was rated on a 4-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). Higher scores indicated a higher level of mircroaggression.
Change from Baseline Social Distance from People with Mental Illness within 10 minutes post-experiment, and at 1-week follow-up | baseline, within 10 minutes post-experiment, and 1-week follow-up
  The 8-item Social Distancing Scale was used to measure the social distance from people with mental illnesses. Each item was rated on a 6-point Likert scale from 1 (very willing) to 6 (very unwilling). Higher scores indicated a higher level of social distance from people with mental illness.
Perceived autonomy | within 10 minutes post-experiment
  To assess perceived autonomy of the Web page experience, the 10-item Self Determination Scale (SDS) was used in the post-experiment questionnaire. Each item was a pair of opposite statements, where participants rated their level of perceived choice and self-awareness with a slider from 1 (only A feels true) to 5 (only B feels true). Higher scores indicated a higher level of perceived autonomy.
Immersiveness | within 10 minutes post-experiment
  The 15-item Transportation Scale was used to assess participants' immersiveness in the Web experience. It had a 4-point Likert scale from 1 (very much) to 4 (not at all). Items 2, 5 and 9 were framed negatively. All the items are scored in the direction that higher scores indicated a higher level of immersivenss.

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Wing-Sze Mak, PhD, Study Chair — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The identifiable personal information collected will be de-linked from the research data and stored separately. The research data will receive a unique number that cannot be traced back to the individuals.
  All information obtained in the course of this experiment will be used for research purposes only; it will be protected and kept confidential by the researchers of this project and not be shared with a third party unless forced by law.
  The identifiable information will be destroyed after data analysis and reporting.

REFERENCES:
- [Derived] Fong THC, Mak WWS. The Effects of Internet-Based Storytelling Programs (Amazing Adventure Against Stigma) in Reducing Mental Illness Stigma With Mediation by Interactivity and Stigma Content: Randomized Controlled Trial. J Med Internet Res. 2022 Aug 12;24(8):e37973. doi: 10.2196/37973. PMID 35969460
- See also: Related Info — https://antistigma.psy.cuhk.edu.hk/